CLINICAL TRIAL: NCT04735497
Title: Patient Ventilator Asynchrony as a Predictor of Weaning Failure in Mechanically Ventilated COPD Patients
Brief Title: Ventilator Asynchrony as a Predictor of Weaning Failure
Status: Completed | Type: Observational
Sponsor: Reham Mohammed Elmorshedy (Other)
Responsible Party: Sponsor-Investigator, Reham Mohammed Elmorshedy, Lecturer, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Ventilator Asynchrony
Record Dates: First submitted 2021-01-11; First posted 2021-02-03 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Chronic Obstructive Pulmonary Disease(COPD)
Keywords: mechanically ventilated; weaning failure; COPD; asynchrony
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Failed Weaning: Patients who failed to be liberated from mechanical ventillation
- Successful Weaning: Patients who were liberated from mechanical ventillation and needed no respiratory support

SUMMARY:
Patient ventilator asynchrony is a common problem in mechanically ventilated patients .It is associated with adverse effects including increased work of breathing, patient discomfort, increased need for sedation, prolonged mechanical ventilation , weaning difficulties and weaning failure. 100 mechanically ventilated COPD patients were enrolled in this prospective study .Detection of patient ventilator asynchrony was done on 30-minute sessions at 12, 24, 36, and 48 hours following intubation by visual assessment of pressure, flow and volume graphs on ventilator .

DETAILED DESCRIPTION:
Patient-ventilator asynchrony is defined as a lack of organization between the patient and ventilator timing of both inspiration and expiration . It is a commonly reported problem during mechanical ventilation. Thille et al. found that 24% of patients developed asynchrony in at least ten percent of their breaths, moreover they stated that the most frequent asynchronies was each of ineffective triggering and double triggering . Eighty percent of chronic obstructive pulmonary disease (COPD) patients experienced ineffective triggering, where it is considered the most frequent asynchrony in this group of patients. Asynchrony between Patient and ventilator also leads to prolonged duration of invasive ventilation, and increase possibility of weaning failure.

Both spread and intensity of asynchrony during the early phase of weaning in COPD patients has never satisfactorily described. The aim of the current study was to describe the patient-ventilator asynchrony and its impact on weaning outcome in mechanically ventilated COPD patients.

ELIGIBILITY:
Inclusion Criteria:

All COPD patients who were diagnosed after history ,physical examination radiology and pulmonary function tests and required mechanical ventilation.

Exclusion Criteria:

1. Age < 18 years
2. Tracheostomy
3. Failure to trigger breaths even in cases of receiving neuromuscular blocking agents.
4. Encephalopathy which is not caused by hypercapnia or hypoxemia either post arrest or due to cerebrovascular stroke
5. Patients with unplanned weaning
6. COPD patients where intubation not related to exacerbation e.g. acute pulmonary edema.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All COPD patients who were diagnosed after history ,physical examination ,radiology and pulmonary function tests and required mechanical ventilation.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
To study effect of different types of ventilator asynchrony on weaning in mechanically ventilated COPD patients | One year
  Detection of patient ventilator asynchrony was done on 30-minute sessions following intubation by visual assessment of pressure, flow
  and volume graphs on ventilator .Repeated measures are done from the begining of mechanical ventilation and type of asynchronies including ineffective trigger double trigger, auto trigger , delayed cycle, early cycle and flow asynchrony. were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Samiaa Sadek, Ass.Lecturer, Principal Investigator — Assiut University
Locations (1):
- Assuit University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No